CLINICAL TRIAL: NCT06429410
Title: Effects of Daily Supplementation With Milk Powder on Body Composition and Physical Performance in Middle-aged and Older Adults: A Randomized Control Trial
Brief Title: Effects of Milk Powder Intervention on Body Composition and Physical Performance in Middle-aged and Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MN-2024-04
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- fortified formula milk powder group (Experimental): Fortified formula milk powder is supplemented with whey protein, calcium, vitamin D, colostrum basic protein, β-hydroxy-β-methylbutyrate, and sodium hyaluronate, and packaged in 25-gram sachets. The milk powder is consumed orally, two sachets per day, for a duration of 24 weeks.
  Interventions: Dietary Supplement: fortified formula milk powder
- formula milk powder group (Experimental): Formula milk powder is supplemented with whey protein, calcium, vitamin D, colostrum basic protein, and sodium hyaluronate, and packaged in 25-gram sachets. The milk powder is consumed orally, two sachets per day, for a duration of 24 weeks.
  Interventions: Dietary Supplement: formula milk powder
- regular milk powder group (Placebo Comparator): Regular milk powder does not contain and additional supplementation, and the color, flavor, shape, taste, and weight are same with the formula milk powder.
  Interventions: Dietary Supplement: regular milk powder
- observation group (No Intervention): Participants in the observation group did not receive any supplementation.

INTERVENTIONS:
Dietary Supplement: fortified formula milk powder — Fortified formula milk powder supplemented with whey protein, calcium, vitamin D, colostrum basic protein, β-hydroxy-β-methylbutyrate, and sodium hyaluronate per day orally for 24 weeks.
  Arms: fortified formula milk powder group
Dietary Supplement: formula milk powder — Formula milk powder supplemented with whey protein, calcium, vitamin D, colostrum basic protein, and sodium hyaluronate per day orally for 24 weeks.
  Arms: formula milk powder group
Dietary Supplement: regular milk powder — Regular milk powder does not contain and additional supplementation, and the color, flavor, shape, taste, and weight are same with the formula milk powder.
  Arms: regular milk powder group

SUMMARY:
This study aims to conduct a 24-week intervention involving formula milk powder for middle-aged and elderly individuals, assessing its impact on body composition and physical performance in comparison to interventions using regular milk powder and individuals without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years old and older;
* BMI <22kg/m2;
* Calf circumference <33cm in women or <34cm in men, or SARC-F ≥ 4, or SARC-Claf ≥ 11;
* Living in Guangzhou and having no plan to move in the next 6 months;
* Willing to participate in the study.

Exclusion Criteria:

* Lactose intolerance;
* Complicated with severe diseases;
* Unable to conduct study procedures;
* Participating in any other intervention studies.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
lean body mass | up to 24 weeks
  At baseline, and 24 weeks, investigators will use DXA to examine lean body mass and fat composition.

SECONDARY OUTCOMES:
cardiorespiratory fitness | up to 24 weeks
  At baseline, and 24 weeks, investigators will use cardiopulmonary exercise testing (CPET) on a cycle ergometer to evaluate cardiorespiratory fitness.
muscle strength | up to 24 weeks
  At baseline, 12, and 24 weeks, investigators will test hand grip to assess muscle strength.
physical performance | up to 24 weeks
  At baseline, 12, and 24 weeks, investigators will test the Short Physical Performance Battery (SPPB) to assess muscular function.
the levels of blood metabolic markers for bone and muscle | up to 24 weeks
  At baseline, and 24 weeks, blood samples will be drawn and serum indexes of bone and muscle metabolism will be test, including myostatin, PINP, CTx, and osteocalcin.